CLINICAL TRIAL: NCT00588107
Title: Partnership for Health: A Web-Based Smoking Intervention For Cancer Survivors
Brief Title: A Web Site and Print Materials Intervention for Smoking Intervention for Childhood and Young Adult Cancer Survivors
Acronym: PFH2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); St. Jude Children's Research Hospital (Other); Princess Margaret Hospital, Canada (Other); The Hospital for Sick Children (Other); University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Karen Emmons, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 05-032; R01CA106914 (NIH)
Record Dates: First submitted 2007-12-24; First posted 2008-01-08 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Cancer
Keywords: Cancer; Smoker; Web based intervention; Partnership for Health; Cancer Survivors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web site access (Experimental): Web intervention- and access to pharmacotherapy
  Interventions: Other: Web Intervention
- print materials (Active Comparator): Receives tailored print materials and access to pharmacotherapy (Materials condition)
  Interventions: Behavioral: print materials

INTERVENTIONS:
Other: Web Intervention — Receives pharmacotherapy and access to an interactive Web site (Web condition). The Web site will offer tailored intervention messages and strategies in an interactive format that is much less labor-intensive and costly than the prior PFH peer telephone counseling intervention.
  Arms: Web site access
Behavioral: print materials — tailored print materials designed to aid in smoking reduction and cessation
  Arms: print materials

SUMMARY:
The purpose of this study was to compare two different ways of helping people who have had childhood cancer, leukemia, tumors or similar illnesses learn health information and information about trying to quit smoking. All participants received materials in the mail about their health, survivorship, and smoking. Some participants were also invited to use a website. The goal of the study was to see which is a better way to get information about health issues, survivorship, and smoking.

DETAILED DESCRIPTION:
The study was a randomized controlled trial with two groups. It was designed to demonstrate the efficacy and cost-effectiveness of a Web-based format of the PFH intervention, compared to a written Materials control condition. The study was conducted among childhood and young adult cancer survivors, who smoke, at four survivor clinics. Participants in both conditions received access to pharmacotherapy at no cost. Participants in the Web condition received access to an interactive Web site that focuses on survivorship, health, and smoking.

Participants in the Web condition received access to an interactive Web site that focuses on survivorship, health, and smoking. Participants in the Materials control group received tailored and targeted print materials.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with cancer before age 35
* Currently be ≥ 18 years of age and ≤ 55 years of age
* 2 or more years out of cancer treatment
* Be mentally capable of providing informed consent
* Be reachable by telephone for screening and survey completion
* Be a current smoker (defined as having taken one puff of a cigarette in the last 30 days)
* Fluent in English

Exclusion Criteria:

* Currently undergoing active treatment for cancer

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 374 (Actual)
Dates: Start 2005-09; Primary Completion 2010-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome is smoking cessation | 15 months post BL

SECONDARY OUTCOMES:
Secondary outcome: cost-effectiveness, intervention dose delivered, reach, impact, quit attempts, motivation to quit, and use of pharmacotherapy | 15 months post BL

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Emmons, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- DFCI, Boston, Massachusetts, United States

REFERENCES:
- [Background] de Moor JS, Puleo E, Ford JS, Greenberg M, Hodgson DC, Tyc VL, Ostroff J, Diller LR, Levy AG, Sprunck-Harrild K, Emmons KM. Disseminating a smoking cessation intervention to childhood and young adult cancer survivors: baseline characteristics and study design of the partnership for health-2 study. BMC Cancer. 2011 May 11;11:165. doi: 10.1186/1471-2407-11-165. PMID 21569345
- [Background] Nagler RH, Puleo E, Sprunck-Harrild K, Emmons KM. Internet use among childhood and young adult cancer survivors who smoke: implications for cessation interventions. Cancer Causes Control. 2012 Apr;23(4):647-52. doi: 10.1007/s10552-012-9926-9. Epub 2012 Feb 28. PMID 22370697
- [Background] Tyc VL, Puleo E, Emmons K, de Moor JS, Ford JS. Smoking Restrictions Among Households of Childhood and Young Adult Cancer Survivors: Implications for Tobacco Control Efforts. J Adolesc Young Adult Oncol. 2013 Mar;2(1):17-24. doi: 10.1089/jayao.2012.0019. PMID 23610739
- [Background] Nagler RH, Puleo E, Sprunck-Harrild K, Viswanath K, Emmons KM. Health media use among childhood and young adult cancer survivors who smoke. Support Care Cancer. 2014 Sep;22(9):2497-507. doi: 10.1007/s00520-014-2236-x. Epub 2014 Apr 13. PMID 24728617
- [Background] Ford JS, Puleo E, Sprunck-Harrild K, deMoor J, Emmons KM. Perceptions of risk among childhood and young adult cancer survivors who smoke. Support Care Cancer. 2014 Aug;22(8):2207-17. doi: 10.1007/s00520-014-2165-8. PMID 24659242
- [Result] Emmons KM, Sprunck-Harrild K, Puleo E, de Moor J. Provider advice about smoking cessation and pharmacotherapy among cancer survivors who smoke: practice guidelines are not translating. Transl Behav Med. 2013 Jun;3(2):211-7. doi: 10.1007/s13142-013-0202-7. PMID 23894256
- [Result] Emmons KM, Puleo E, Sprunck-Harrild K, Ford J, Ostroff JS, Hodgson D, Greenberg M, Diller L, de Moor J, Tyc V. Partnership for health-2, a web-based versus print smoking cessation intervention for childhood and young adult cancer survivors: randomized comparative effectiveness study. J Med Internet Res. 2013 Nov 5;15(11):e218. doi: 10.2196/jmir.2533. PMID 24195867